CLINICAL TRIAL: NCT05693337
Title: Infrared (FLIR) Imaging as a Monitor for Sympathetic Blocks in Complex Regional Pain Syndrome (CRPS)
Brief Title: Infrared Imaging in Complex Regional Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1996
Record Dates: First submitted 2022-09-09; First posted 2023-01-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Complex Regional Pain Syndromes
Keywords: complex; regional; pain; FLIR; Sympathetic Block
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- FLIR Imaging: All patients recruited for this study will receive FLIR imaging to monitor the success of a lumbar sympathetic block for CRPS
  Interventions: Device: Forward Looking Infrared Radar (FLIR) thermal imaging

INTERVENTIONS:
Device: Forward Looking Infrared Radar (FLIR) thermal imaging — The FLIR camera will collect temperature recordings pre-procedure and 5 minutes post-procedure, which will be used to calculate a delta T to assess achievement of a successful sympathetic block.

SUMMARY:
This research proposal aims to investigate the potential use of Infrared (FLIR) imaging to monitor the successful achievement of the sympathetic blockade in patients with complex regional pain syndrome (CRPS).

DETAILED DESCRIPTION:
Sympathetic blocks are clinically used to diagnose and treat sympathetically mediated pain. Despite the frequent use of these blocks, there remains a need for an objective method to determine the achievement of a sympathetic block in the clinical setting.

Current clinical practice assess the success of a sympathetic block by observation of clinical signs of sympathetic blockade. These signs include monitoring skin temperature, pulse amplitude, blood oxygen, or any combination of these methods. However, clinical signs of sympathetic blockade often demonstrate an unpredictable or delayed response and can make monitoring difficult.

Therefore, it is necessary to develop an objective monitoring method that is reliable, rapid response, and not affected by the other confounders. One potential method is the use of thermal camera imaging (FLIR).

Such a monitor could increase procedural accuracy and efficiency, thus improving patient care. To plan the prospective treatment options, objective confirmation of successful sympathetic block is essential to differentiate sympathetically mediated pain (SMP) versus sympathetically independent pain (SIP).

In this context, utilization of a monitor with a rapid response and easy clinical applicability, would serve as an objective endpoint for evaluating sympathetic blockade both clinically and for future research.

Therefore, this research proposal aims to investigate the infrared (FLIR) thermal camera as an objective method for determining the achievement of sympathetic block in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 85 years old
* Providing CRPS diagnostic criteria by using Budapest Clinical criteria [16]
* The patient has had pain and other symptoms for more than 3 months
* Not responding to conventional medical treatments and multidisciplinary approach
* High NRS detection in pain assessment despite appropriate treatment (NRS = and > 6/10).
* Pain is a limitation in the patient's functional capacity despite appropriate treatment.

Exclusion Criteria:

* Patients with suspected disc herniation, spinal stenosis, myelopathy, and suspected radiculopathy in detailed examinations and examinations (MRI, CT).
* Systemic or local infection
* Coagulation disorders
* History of allergy to contrast material
* Malignancy
* Pregnancy
* Uncontrollable medical and psychiatric condition
* The patients diagnosed with dysautonomia, sympathetic dysfunction (such as Raynaud disease or Buerger disease), sweating disorders (such as acquired idiopathic generalized anhidrosis), and patients on vasoactive drugs, the mechanism of action is directly on the vascular tone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed to be implemented in a single center in an academic pain center that is specialized in musculoskeletal pain. In a pain center with a high experience in clinical and academic fields, it is planned to apply lumbar sympathetic blocks to the patients diagnosed with CRPS. The Budapest Clinical Diagnostic Criteria will be used to diagnose CRPS Type 1 patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Circulation Improvement | 5 minutes post procedure
  Improvement of circulation and perfusion in the affected limb by FLIR camera in CRPS patients at a 5-minutes time point after the completion of the block.

SECONDARY OUTCOMES:
Comparison between FLIR and Standard Measuring | 5 minutes post procedure
  The developed quantitative measurement will be compared with the "qualitative assessment of clinical signs of sympathectomy" scale at 5-minute post-procedure to determine which method was superior to detecting sympathetic block.
Numerical Pain Score Correlation | 10 days post procedure
  The developed quantitative measurement will be compared with the currently used NRS values at postoperative follow-up (1-2 weeks) time points after completion of the sympathetic block.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, MD, Principal Investigator — Hospital for Special Surgery, Department of Anesthesiology
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers.

REFERENCES:
- [Background] Day M. Sympathetic blocks: the evidence. Pain Pract. 2008 Mar-Apr;8(2):98-109. doi: 10.1111/j.1533-2500.2008.00177.x. PMID 18366465
- [Background] McCormick ZL, Hendrix A, Dayanim D, Clay B, Kirsling A, Harden N. Lumbar Sympathetic Plexus Block as a Treatment for Postamputation Pain: Methodology for a Randomized Controlled Trial. Pain Med. 2018 Dec 1;19(12):2496-2503. doi: 10.1093/pm/pny041. PMID 29528455
- [Background] Krumova EK, Gussone C, Regeniter S, Westermann A, Zenz M, Maier C. Are sympathetic blocks useful for diagnostic purposes? Reg Anesth Pain Med. 2011 Nov-Dec;36(6):560-7. doi: 10.1097/AAP.0b013e318229bbee. PMID 21941221
- [Background] Park SY, Nahm FS, Kim YC, Lee SC, Sim SE, Lee SJ. The cut-off rate of skin temperature change to confirm successful lumbar sympathetic block. J Int Med Res. 2010 Jan-Feb;38(1):266-75. doi: 10.1177/147323001003800131. PMID 20233538
- [Background] Gungor S, Rana B, Fields K, Bae JJ, Mount L, Buschiazzo V, Storm H. Changes in the Skin Conductance Monitor as an End Point for Sympathetic Nerve Blocks. Pain Med. 2017 Nov 1;18(11):2187-2197. doi: 10.1093/pm/pnw318. PMID 28158730
- [Background] Cheng J, Salmasi V, You J, Grille M, Yang D, Mascha EJ, Cheng OT, Zhao F, Rosenquist RW. Outcomes of Sympathetic Blocks in the Management of Complex Regional Pain Syndrome: A Retrospective Cohort Study. Anesthesiology. 2019 Oct;131(4):883-893. doi: 10.1097/ALN.0000000000002899. PMID 31365367
- [Background] Gungor S, Aiyer R, Baykoca B. Sympathetic blocks for the treatment of complex regional pain syndrome: A case series. Medicine (Baltimore). 2018 May;97(19):e0705. doi: 10.1097/MD.0000000000010705. PMID 29742728
- [Background] Gungor S, Aiyer R. Extrapyramidal signs occurring after sympathetic block for complex regional pain syndrome responding to diphenhydramine: Two case reports. Medicine (Baltimore). 2018 Jun;97(26):e11301. doi: 10.1097/MD.0000000000011301. PMID 29953015
- [Background] O'Connell NE, Wand BM, McAuley J, Marston L, Moseley GL. Interventions for treating pain and disability in adults with complex regional pain syndrome. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD009416. doi: 10.1002/14651858.CD009416.pub2. PMID 23633371
- [Background] Ghosh P, Gungor S. Utilization of Concurrent Dorsal Root Ganglion Stimulation and Dorsal Column Spinal Cord Stimulation in Complex Regional Pain Syndrome. Neuromodulation. 2021 Jun;24(4):769-773. doi: 10.1111/ner.13144. Epub 2020 Mar 11. PMID 32162402
- [Background] Noori SA, Gungor S. Spinal epidural abscess associated with an epidural catheter in a woman with complex regional pain syndrome and selective IgG3 deficiency: A case report. Medicine (Baltimore). 2018 Dec;97(50):e13272. doi: 10.1097/MD.0000000000013272. PMID 30557971
- See also: London: Royal College of Physicians — https://www.rcplondon.ac.uk/guidelines-policy/complex-regional-pain-syndrome-adults